CLINICAL TRIAL: NCT01647347
Title: Effects of Ultrasonic Debridement With PVP-iodine Irrigation on Post-treatment Bacteraemia Compared to Ultrasonic Debridement With Water
Brief Title: PVP Iodine Effect on Post Debridement Bacteraemia
Acronym: PJB 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PJB 1
Record Dates: First submitted 2012-07-16; First posted 2012-07-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Bacteraemia Post Debridement
Keywords: bacteria; bacteremia; PVP-iodine; periodontitis
MeSH Terms: conditions — Bacteremia; Periodontitis | interventions — Povidone-Iodine; Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test treatment (Experimental): Test treatment:
  * 1 min mouthwash with 10% PVP-iodine
  * 1 min subgingival rinsing with 10% PVP-iodine
  * 1 min ultrasonic debridement with 10% PVP-iodine as cooling liquid
  * blood sampling from the V.mediana cupidi
  Interventions: Drug: Supra- and subgingival rinsing with 10% PVP-iodine
- Control group (Placebo Comparator): Control:
  * 1 min mouthwash with water
  * 1 min subgingival rinsing with water
  * 1 min ultrasonic debridement with water as cooling liquid
  * blood sampling from the V.mediana cupidi
  Interventions: Other: Water

INTERVENTIONS:
Drug: Supra- and subgingival rinsing with 10% PVP-iodine — rinsing prior to and during subgingival ultrasonic debridement
  Other Names: Betadine standardized solution (mundipharma, Basel, Switzerland); CH.B. 10070401
  Arms: test treatment
Other: Water
  Arms: Control group

SUMMARY:
The study investigates the effect of supra- and subgingival rinsing of 10% PVP prior to ultrasonic debridement in patients with periodontitis (as compared to rinsing with water) in terms of post treatment bacteraemia.

Study design: Randomized split-mouth (cross-over) study on 20 generally healthy subjects.

DETAILED DESCRIPTION:
Process:

Test treatment:

* 1 min mouthwash with 10% PVP-iodine
* 1 min subgingival rinsing with 10% PVP-iodine
* 1 min ultrasonic debridement with 10% PVP-iodine as cooling liquid
* blood sampling from the V.mediana cupidi

Control:

* 1 min mouthwash with water
* 1 min subgingival rinsing with water
* 1 min ultrasonic debridement with water as cooling liquid
* blood sampling from the V.mediana cupidi

lysis, culturing and analysis of bacteria in the samples

ELIGIBILITY:
Inclusion Criteria:

* generally healthy, adult (≥ 18 years) patients with at least two periodontal pockets of ≥ 5 mm

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy on PVP-iodine
* anticoagulation (exception 100mg/d acetylsalicylic acid)
* high risc for endocarditis
* therapeutical radiation
* participation in other clinical studies
* cognitive impairment (patient unable to understand aim and conduction of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
quantity of bacteraemia in central blood stream | three minutes after starting debridement
  In how many samples a bacterial contamination is found?
quality of bacteraemia in central blood stream | three minutes after starting debridement
  How many CFU are found in each blood sample?

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Sahrmann, Senior Assistant, Principal Investigator — Clinic for Preventive Dentistry, Periodontology and Cariology, University of Zurich
Locations (1):
- Clinic for Preventive Dentistry, Perioodntology and Cariology, University of Zurich, Zurich, Canton of Zurich, Switzerland